CLINICAL TRIAL: NCT00547339
Title: A Phase I and II Study of Stereotactic Body Radiation Therapy (SBRT) for Low and Intermediate Risk Prostate Cancer (SBRT Prostate)
Brief Title: Stereotactic Body Radiation Therapy in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Robert Timmerman, Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCCC-0604122; STU 072010-019; SCCC-062006-010; CDR0000571546 (Registry Identifier: PDQ (Physician Data Query)); UMN-2006UC048; NCT03554369 (obsolete NCT alias)
Record Dates: First submitted 2007-10-19; First posted 2007-10-22 (Estimated); Results first posted 2022-03-24 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery; Clinical Trials, Phase I as Topic; Clinical Trials, Phase II as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Phase 1: Stereotactic Body Radiation Therapy (SBRT) 45 Gy (Experimental): The Phase 1 portion of the study will have a 3+3 design. The dose of SBRT is escalated - 45 Gy
  Interventions: Radiation: stereotactic body radiation therapy (SBRT)- 45 Gy
- Phase 1: Stereotactic Body Radiation Therapy (SBRT)- 47.5 Gy (Experimental): The Phase 1 portion of the study will have a 3+3 design. The dose of SBRT is escalated- 47.5 Gy
  Interventions: Radiation: stereotactic body radiation therapy (SBRT) - 47.5 Gy
- Phase 1: Stereotactic Body Radiation Therapy (SBRT)- 50 Gy (Experimental): The Phase 1 portion of the study will have a 3+3 design. The dose of SBRT is escalated- 50 Gy
  Interventions: Radiation: stereotactic body radiation therapy (SBRT) - 50 Gy (Phase 1)
- Phase 2: Stereotactic Body Radiation Therapy (SBRT)- 50 Gy (Experimental): The dose of SBRT is escalated - 50 Gy in Phase 2
  Interventions: Radiation: stereotactic body radiation therapy (SBRT) - 50 Gy (Phase 2)

INTERVENTIONS:
Radiation: stereotactic body radiation therapy (SBRT)- 45 Gy — Dose of SBRT - 45 Gray (Gy) in five fractions
  Arms: Phase 1: Stereotactic Body Radiation Therapy (SBRT) 45 Gy
Radiation: stereotactic body radiation therapy (SBRT) - 47.5 Gy — Dose of SBRT - 47.5 Gray (Gy) in five fractions
  Other Names: Dose of SBRT - 47.5 Gy in five fractions
  Arms: Phase 1: Stereotactic Body Radiation Therapy (SBRT)- 47.5 Gy
Radiation: stereotactic body radiation therapy (SBRT) - 50 Gy (Phase 1)
  Other Names: Dose of SBRT - 50 Gray (Gy) in five fractions
  Arms: Phase 1: Stereotactic Body Radiation Therapy (SBRT)- 50 Gy
Radiation: stereotactic body radiation therapy (SBRT) - 50 Gy (Phase 2)
  Other Names: Dose of SBRT - 50 Gray (Gy) in five fractions
  Arms: Phase 2: Stereotactic Body Radiation Therapy (SBRT)- 50 Gy

SUMMARY:
RATIONALE: Stereotactic body radiation therapy may be able to send x-rays directly to the tumor and cause less damage to normal tissue.

PURPOSE: This phase I/II trial is studying the side effects and best dose of stereotactic body radiation therapy and to see how well it works in treating patients with prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To escalate the dose of stereotactic body radiotherapy (SBRT) to a tumoricidal dose without exceeding the maximum tolerated dose in patients with organ-confined prostate cancer. (Phase I)
* To determine the late, severe grade 3-5 genitourinary and gastrointestinal toxicity occurring between 270-540 days (i.e., 9-18 months) from the start of the protocol treatment as assessed by CTCAE v3.0. (Phase II)

Secondary

* To determine the dose-limiting toxicity of SBRT in these patients. (Phase I)
* To determine the 2-year biochemical (PSA) control (freedom from PSA failure), disease-free and overall survival, local control, freedom from distant metastases, and the incidence of high-grade adverse events of any type in patients treated with this therapy in order to determine if the therapy is promising enough for further clinical investigation. (Phase II)

OUTLINE: This is a multicenter, phase I dose-escalation study followed by a phase II open-label study.

* Phase I: Patients undergo 5 treatments of stereotactic body radiotherapy (SBRT).
* Phase II: Patients undergo SBRT at the maximum tolerated dose as in phase I. After completion of study treatment, patients are followed at 1.5, 3, 6, 9, and 12 months, every 6 months for 5 years, and then once a year for years 5-10.

PROJECTED ACCRUAL: A total of 97 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * Stage T1a, T1b, T1c disease
  * Stage T2a or T2b
* No direct evidence of regional or distant metastases
* No T2c, T3, or T4 tumors
* Gleason score ≤ 7
* Must meet the following criteria:

  * Prostate-specific antigen (PSA) ≤ 20 ng/mL prior to starting hormonal therapy (if given) for patients with a Gleason score of 2-6
  * PSA ≤ 15 ng/mL prior to starting hormonal therapy (if given) for patients with a Gleason score of 7
  * Risk of pelvic lymph node involvement < 20% according to Roach formula
* Ultrasound-based volume estimation of the prostate gland ≤ 60 g

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-2
* Fertile patients must use effective contraception
* No prior invasive malignancy, except for nonmelanoma skin cancer, unless disease-free for a minimum of 3 years (e.g., carcinoma in situ of the breast, oral cavity, or cervix are allowed)
* No significant urinary obstructive symptoms

  * American Urological Association (AUA) score of ≤ 15 (alpha blockers allowed)
* No history of inflammatory colitis (including Crohn disease and ulcerative colitis)
* No history of significant psychiatric illness
* No severe, active comorbidity including any of the following:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the past 6 months
  * Transmural myocardial infarction within the past 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days prior to registration
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects

    * Laboratory tests for liver function and coagulation parameters are not required for entry into this protocol
  * AIDS (based on current CDC definition) or other immunocompromising condition

    * HIV testing is not required for entry into this protocol

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 9 months since prior hormonal therapy as neoadjuvant therapy or to downsize the prostate gland
* No prior pelvic radiotherapy
* No prior chemotherapy or surgery for prostate cancer
* No prior transurethral resection of the prostate (TURP) or cryotherapy to the prostate
* No plans for other concurrent post-treatment, adjuvant, antineoplastic therapy including surgery, cryotherapy, conventionally fractionated radiotherapy, hormonal therapy, or chemotherapy as part of the treatment for prostate cancer

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2006-07 (Actual); Primary Completion 2014-07-20 (Actual); Study Completion 2022-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert D. Timmerman, MD, Study Chair — Simmons Cancer Center
Locations (5):
- United States (5):
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - MD Anderson Cancer Center Orlando Florida, Orlando, Florida
  - University of Minnesota Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Prairie Lakes Cancer Center, Watertown, South Dakota
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 94 patients were recruited. Two patients withdrew consent before treatment and an additional patient had Gleason 9 disease upon pathology review and was excluded from the analysis. A total of 91 patients were analyzed.
Groups:
- Phase 1: Dose Escalation 45 Gy Arm: Dose escalation portion will be 9 Gy per fraction for 5 fractions (total dose = 45 Gy).
- Phase 1: Dose Escalation 47.5 Gy Arm: Dose escalation portion will be 9.5 Gy per fraction for 5 fractions (total dose = 47.5 Gy).
- Phase 1: Dose Escalation 50 Gy Arm; Phase 2: Dose Escalation 50 Gy Arm: Dose escalation portion will be 9 Gy per fraction for 5 fractions (total dose = 50 Gy).
Period: Overall Study
Arm/Group | Phase 1: Dose Escalation 45 Gy Arm | Phase 1: Dose Escalation 47.5 Gy Arm | Phase 1: Dose Escalation 50 Gy Arm | Phase 2: Dose Escalation 50 Gy Arm
Started | 15 | 15 | 15 | 47
Completed | 15 | 15 | 14 | 47
Not Completed | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: A total of 94 patients were recruited. Two patients withdrew consent before treatment and an additional patient had Gleason 9 disease upon pathology review and was excluded from the analysis. A total of 91 patients were analyzed.
Groups:
- Phase 1: SBRT- 45 Gy(SBRT) 45 Gy.: The dose of Stereotactic Body Radiation Therapy (SBRT) is - 45 Gy in Phase 1
- Phase 1: SBRT- 47.5 Gy: The dose of Stereotactic Body Radiation Therapy (SBRT) is - 47.5 Gy in Phase 1
- Phase 1: Stereotactic Body Radiation Therapy (SBRT) 50 Gy.: The dose of Stereotactic Body Radiation Therapy (SBRT) is - 50 Gy in Phase 1
- Phase 2: Stereotactic Body Radiation Therapy (SBRT)- 50 Gy: The dose of SBRT is escalated- 50 Gy in Phase 2 stereotactic body radiation therapy (SBRT) - 50 Gy (Phase 2).
- Total: Total of all reporting groups
Arm/Group | Phase 1: SBRT- 45 Gy(SBRT) 45 Gy. | Phase 1: SBRT- 47.5 Gy | Phase 1: Stereotactic Body Radiation Therapy (SBRT) 50 Gy. | Phase 2: Stereotactic Body Radiation Therapy (SBRT)- 50 Gy | Total
Number analyzed (Participants) | 15 | 15 | 14 | 47 | 91
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 67 [55 to 82] | 67 [58 to 76] | 67 [53 to 78] | 65 [52 to 80] | 66 [53 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 15 | 15 | 14 | 47 | 91
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 9 | 13 | 12 | 32 | 66
  Non-White | 6 | 2 | 2 | 15 | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicity (Phase 1 Only)
Description: Dose-limiting toxicity (DLT) was defined as grade 3 to 5 GI, genito urinary, sexual, or neurologic toxicity attributed to therapy occurring within 90 days of registration using Common Terminology Criteria of Adverse Events(version 3)
Time Frame: 90 days after start of treatment
Population: Total enrolled was 47 patients to the phase I study, although two withdrew consent before treatment and an additional patient had Gleason 9 disease upon pathology and was excluded from the analysis. MTD not met in Phase I.
Measure: Number; unit: participants
Groups:
- Phase 1: SBRT- 45 Gy: The dose of Stereotactic Body Radiation Therapy (SBRT) is - 45 Gy in Phase 1
- Phase 1: SBRT- 50 Gy: The dose of Stereotactic Body Radiation Therapy (SBRT) is - 50 Gy in Phase 1
Arm/Group | Phase 1: SBRT- 45 Gy | Phase 1: SBRT- 47.5 Gy | Phase 1: SBRT- 50 Gy | Phase 2: Stereotactic Body Radiation Therapy (SBRT)- 50 Gy
Number analyzed (Participants) | 15 | 15 | 14 | 47
participants | 0 | 0 | 0 | 0

2. Primary Outcome: No. of Late Severe GU Toxicity (for Phase 2 Only)
Description: To determine late severe GU toxicity defined as grade 3-5 occurring between 279-540 days (i.e., 9-18 months) from the start of protocol treatment. Toxicity was defined using the National Cancer Institute Common Toxicity Criteria for Adverse Events (CTCAE) v.3.0. CTCAE uses a range of grades from 1 to 5; 1 - Mild 2 - Moderate 3 - Severe 4 - Life-threatening 5 - Death.
Time Frame: 18 months
Measure: Number; unit: participants
Arm/Group | Phase 2: Stereotactic Body Radiation Therapy (SBRT)- 50 Gy
Number analyzed (Participants) | 47
participants
  Grade III | 3
  Grade IV | 1
  Grade V | 0

3. Primary Outcome: No. of Late Severe GI Toxicity (for Phase 2 Only)
Description: To determine late severe GI toxicity defined as grade 3-5 occurring between 279-540 days (i.e., 9-18 months) from the start of protocol treatment. Toxicity was defined using the National Cancer Institute Common Toxicity Criteria for Adverse Events (CTCAE) v.3.0. CTCAE uses a range of grades from 1 to 5; 1 - Mild 2 - Moderate 3 - Severe 4 - Life-threatening 5 - Death.
Time Frame: 18 months
Measure: Number; unit: participants
Arm/Group | Phase 2: Stereotactic Body Radiation Therapy (SBRT)- 50 Gy
Number analyzed (Participants) | 47
participants
  Grade III | 4
  Grade IV | 2
  Grade V | 0

4. Secondary Outcome: GU Toxicity (Only Phase 2)
Description: To determine acute severe GU toxicity is defined as grade 3-5 occurring prior to 270 days from the start of the protocol treatment. Toxicity was defined using the National Cancer Institute Common Toxicity Criteria for Adverse Events (CTCAE) v.3.0. CTCAE uses a range of grades from 1 to 5; 1 - Mild 2 - Moderate 3 - Severe 4 - Life-threatening 5 - Death.
Time Frame: 9 months from start of treatment
Measure: Number; unit: participants
Arm/Group | Phase 2: Stereotactic Body Radiation Therapy (SBRT)- 50 Gy
Number analyzed (Participants) | 47
participants
  Grade III | 0
  Grade IV | 0
  Grade V | 0

5. Secondary Outcome: GI Toxicity
Description: To determine acute severe GI toxicity is defined as grade 3-5 occurring prior to 270 days from the start of the protocol treatment. Toxicity was defined using the National Cancer Institute Common Toxicity Criteria for Adverse Events (CTCAE) v.3.0. CTCAE uses a range of grades from 1 to 5; 1 - Mild 2 - Moderate 3 - Severe 4 - Life-threatening 5 - Death.
Time Frame: 9 months from start of treatment
Measure: Number; unit: participants
Arm/Group | Phase 2: Stereotactic Body Radiation Therapy (SBRT)- 50 Gy
Number analyzed (Participants) | 47
participants
  Grade III | 1
  Grade IV | 1
  Grade V | 0

6. Secondary Outcome: Non-GU Toxicity
Description: To determine non-GU (genitourinary) toxicity is defined as grade 3-5. Toxicity was defined using the National Cancer Institute Common Toxicity Criteria for Adverse Events (CTCAE) v.3.0. CTCAE uses a range of grades from 1 to 5; 1 - Mild 2 - Moderate 3 - Severe 4 - Life-threatening 5 - Death.
Time Frame: 60 months
Population: The data was not collected.
Groups:
- Phase 1: Stereotactic Body Radiation Therapy (SBRT)- 50 Gy: The dose of Stereotactic Body Radiation Therapy (SBRT) is - 50 Gy in Phase 1
Arm/Group | Phase 1: SBRT- 45 Gy | Phase 1: SBRT- 47.5 Gy | Phase 1: Stereotactic Body Radiation Therapy (SBRT)- 50 Gy | Phase 2: Stereotactic Body Radiation Therapy (SBRT)- 50 Gy
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Non-GI Toxicity
Description: To determine non-GI (gastrointestinal) toxicity is defined as grade 3-5. Toxicity was defined using the National Cancer Institute Common Toxicity Criteria for Adverse Events (CTCAE) v.3.0. CTCAE uses a range of grades from 1 to 5; 1 - Mild 2 - Moderate 3 - Severe 4 - Life-threatening 5 - Death.
Time Frame: 60 months
Population: The data was not collected.
Arm/Group | Phase 1: SBRT- 45 Gy | Phase 1: SBRT- 47.5 Gy | Phase 1: Stereotactic Body Radiation Therapy (SBRT)- 50 Gy | Phase 2: Stereotactic Body Radiation Therapy (SBRT)- 50 Gy
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Freedom From Biochemical Failure
Description: Biochemical failure RTOG (Radiation Therapy Oncology Group)-ASTRO (American Society for Therapeutic Radiology and Oncology) definition (also known as Phoenix definition). Thus, when the PSA rises by more than 2 ng/ml above the lowest level (nadir) achieved after treatment, biochemical failure has occurred and the date of the failure is recorded at the time the nadir plus 2 ng/ml level is reached.
Time Frame: 36 months
Population: Phase 1: SBRT- 45Gy was the only arm to have a patient with biochemical progression.
Measure: Number; unit: percentage of participants
Groups:
- Phase 1: SBRT - 45 Gy: The dose of Stereotactic Body Radiation Therapy (SBRT) is - 45 Gy in Phase 1
- Phase 1: SBRT- 47.5 Gy: The dose of Stereotactic Body Radiation Therapy (SBRT) is escalated to 47.5 Gy in Phase 1
- Phase 1: SBRT- 50 Gy: The dose of Stereotactic Body Radiation Therapy (SBRT) is escalated to 50 Gy in Phase 1
- Phase 2: SBRT - 50 Gy: The dose of Stereotactic Body Radiation Therapy (SBRT) is escalated to 50 Gy in Phase 2
Arm/Group | Phase 1: SBRT - 45 Gy | Phase 1: SBRT- 47.5 Gy | Phase 1: SBRT- 50 Gy | Phase 2: SBRT - 50 Gy
Number analyzed (Participants) | 15 | 15 | 14 | 47
percentage of participants | 90.9 | 100 | 100 | 100

9. Secondary Outcome: Overall Survival
Description: The survival time will be measured from the date of accession to the date of death.
Time Frame: 60 months
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1: SBRT- 45 Gy | Phase 1: SBRT- 47.5 Gy | Phase 1: SBRT- 50 Gy | Phase 2: Stereotactic Body Radiation Therapy (SBRT)- 50 Gy
Number analyzed (Participants) | 15 | 15 | 14 | 47
percentage of participants | 71.5 | 85 | 92 | 98

10. Secondary Outcome: Disease Specific Survival
Description: Disease-Specific Survival Disease-specific survival will be measured from the date of study entry to the date of death due to prostate cancer as the percentage of participants who survived the prostrate cancer disease.
Time Frame: 60 months
Measure: Number; unit: percentage of participants
Groups:
- Phase 2: SBRT- 50 Gy: The dose of SBRT is escalated- 50 Gy in Phase 2 stereotactic body radiation therapy (SBRT) - 50 Gy (Phase 2).
Arm/Group | Phase 1: SBRT- 45 Gy | Phase 1: SBRT- 47.5 Gy | Phase 1: SBRT- 50 Gy | Phase 2: SBRT- 50 Gy
Number analyzed (Participants) | 15 | 15 | 14 | 47
percentage of participants | 100 | 100 | 100 | 100

11. Secondary Outcome: Clinical Progression Including Local/Regional and Distant Relapse
Description: Clinical progression including local/regional and distant relapse is measured using Kaplan-Meier method
Time Frame: 60 months
Measure: Number; unit: number of participants
Groups:
- Phase 2: SBRT - 50 Gy: The dose of Stereotactic Body Radiation Therapy (SBRT) is escalated - 50 Gy in Phase 2
Arm/Group | Phase 1: SBRT - 45 Gy | Phase 1: SBRT- 47.5 Gy | Phase 1: SBRT- 50 Gy | Phase 2: SBRT - 50 Gy
Number analyzed (Participants) | 15 | 15 | 14 | 47
number of participants | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 60 months
Arm/Group | Phase 1: SBRT- 45 Gy | Phase 1: SBRT- 47.5 Gy | Phase 1: SBRT- 50 Gy | Phase 2: Stereotactic Body Radiation Therapy (SBRT)- 50 Gy
All-Cause Mortality (participants affected / at risk) | 4/15 | 2/15 | 1/14 | 1/47
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/14 | 0/47
Other Adverse Events (participants affected / at risk) | 8/15 | 8/15 | 11/14 | 33/47
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: SBRT- 45 Gy (N=15) | Phase 1: SBRT- 47.5 Gy (N=15) | Phase 1: SBRT- 50 Gy (N=14) | Phase 2: Stereotactic Body Radiation Therapy (SBRT)- 50 Gy (N=47)
Urinary Frequency (Renal and urinary disorders) | 4 | 5 | 8 | 5 — Non-Sexual Domain
Urinary Urgency (Renal and urinary disorders) | 3 | 3 | 1 | 0 — Non-Sexual Domain
Cystitis (Renal and urinary disorders) | 3 | 1 | 2 | 2 — Non-Sexual Domain
Urinary Incontinence (Renal and urinary disorders) | 1 | 3 | 0 | 1 — Non-Sexual Domain
Hematuria (Renal and urinary disorders) | 2 | 0 | 1 | 1 — Non-Sexual Domain
Urinary Retention (Renal and urinary disorders) | 1 | 0 | 0 | 1 — Non-Sexual Domain
Dysuria (Renal and urinary disorders) | 0 | 1 | 1 | 4 — Non-Sexual Domain
Bladder Ulcer (Renal and urinary disorders) | 0 | 0 | 1 | 0 — Non-Sexual Domain
Urethral Stricture (Renal and urinary disorders) | 0 | 0 | 1 | 0 — Non-Sexual Domain
Rectal Toxicity (Gastrointestinal disorders) | 8 | 8 | 11 | 33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-11-20): https://cdn.clinicaltrials.gov/large-docs/39/NCT00547339/Prot_SAP_000.pdf